CLINICAL TRIAL: NCT06290479
Title: A Three-Group Study to Examine the Efficacy of the Air up® Drinking System at Improving Hydration and Associated Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: air up GmbH (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 20358
Record Dates: First submitted 2024-02-20; First posted 2024-03-04 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Water Intake
Keywords: Hydration; Drinking habits; Flavored water

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Intervention Model: Parallel Assignment Masking: Triple (Participant, Care Provider, Investigator)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking: Triple (Participant, Care Provider, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Air Up® Peach Pod (Experimental): Participants in this arm will use the air up® drinking system with a peach-flavored pod. The intervention aims to test if the flavored scent encourages increased water intake, which will be assessed by self-reported questionnaires and hydration-related health outcomes over 12 weeks.
  Interventions: Dietary Supplement: Air Up® Peach Pod
- Air Up® Orangeade Pod (Experimental): Participants in this arm will use the air up® drinking system with an orangeade-flavored pod. Similar to Arm 1, the intervention will assess the impact of the flavored scent on water consumption and health outcomes, using the same methods of evaluation.
  Interventions: Dietary Supplement: Air Up® Orangeade Pod
- Control - Unscented Pod (No Intervention): Participants in this control arm will use the air up® drinking system with an unscented pod. This group will serve as the control to evaluate the effectiveness of the scented pods in comparison to a baseline with no added scent.

INTERVENTIONS:
Dietary Supplement: Air Up® Peach Pod — Participants in this arm will use the air up® drinking system with a peach-flavored pod.
  Arms: Air Up® Peach Pod
Dietary Supplement: Air Up® Orangeade Pod — Participants in this arm will use the air up® drinking system with an orangeade-flavored pod.
  Arms: Air Up® Orangeade Pod

SUMMARY:
A randomized, controlled trial evaluating the air up® drinking system's impact on hydration and health outcomes. Participants will use air up® with Peach, Orangeade, or unscented pods and their effects on drinking habits, and health outcomes will be assessed over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to use the system
* Generally healthy
* Enjoys the smell of peach or orangeade.

Exclusion Criteria:

* Silicone allergy
* IBS, bariatric surgery,
* pregnancy
* participation in another clinical study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Hydration Habits and Health Outcomes as Measured by the Water Intake Questionnaire and the Hydration-Related Quality of Life Scale | 12 weeks
  This measure evaluates changes in participants' hydration habits and health impacts using questionnaires with a 5-point Likert scale.

SECONDARY OUTCOMES:
Blood Biomarkers | Measured at baseline and at the end of the 12-week study period
  Changes in blood biomarkers (Insulin, HbA1c, and Glucose)

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided